CLINICAL TRIAL: NCT01975259
Title: Investigating the Incretin Effect in Cystic Fibrosis
Acronym: IECF
Status: Completed | Type: Observational
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1004; 2013-003758-26 (EudraCT Number)
Record Dates: First submitted 2013-09-11; First posted 2013-11-04 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glucose Tolerance Test; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; Saline Solution; Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cystic Fibrosis: Adult patients with confirmed cystic fibrosis who are clinically stable. Interventions:
  Oral Glucose Tolerance test (75g 2-hour) Modified Oral Glucose Tolerance Test (50g 4-hours) Matched isoglycemic clamp Hyperglycemic clamp with concurrent GLP-1 infusion Hyperglycemic Clamp with concurrent GIP infusion Hyperglycemic clamp with placebo infusion Liquid Meal Test (Carbohydrate-rich) Continuous Glucose Monitoring
  Interventions: Drug: Oral Glucose Tolerance test (75g 2-hour); Drug: Modified Oral Glucose Tolerance Test (50g 4-hours); Drug: Matched isoglycemic clamp; Drug: Hyperglycemic clamp with concurrent GLP-1 infusion; Drug: Hyperglycemic Clamp with concurrent GIP infusion; Drug: Hyperglycemic clamp with placebo infusion; Other: Liquid Meal Test (Carbohydrate-rich); Other: Liquid Meal Test (Fat-rich); Other: Liquid Meal Test (Mixed); Device: Continuous Glucose Monitoring
- Controls: Adult Non-CF subjects matched for age and body mass index with normal glucose tolerance.
  Oral Glucose Tolerance test (75g 2-hour) Modified Oral Glucose Tolerance Test (50g 4-hours) Matched isoglycemic clamp Hyperglycemic clamp with concurrent GLP-1 infusion Hyperglycemic Clamp with concurrent GIP infusion Hyperglycemic clamp with placebo infusion Liquid Meal Test (Carbohydrate-rich)
  Interventions: Drug: Oral Glucose Tolerance test (75g 2-hour); Drug: Modified Oral Glucose Tolerance Test (50g 4-hours); Drug: Matched isoglycemic clamp; Drug: Hyperglycemic clamp with concurrent GLP-1 infusion; Drug: Hyperglycemic Clamp with concurrent GIP infusion; Drug: Hyperglycemic clamp with placebo infusion; Other: Liquid Meal Test (Carbohydrate-rich); Other: Liquid Meal Test (Fat-rich); Other: Liquid Meal Test (Mixed)

INTERVENTIONS:
Drug: Oral Glucose Tolerance test (75g 2-hour) — A standard 2-hour oral glucose tolerance test where fasted patients (10hours overnight) consume a 75g glucose solution & have glucose levels recorded up to every 30 mins for 2hours
  Other Names: OGTT
Drug: Modified Oral Glucose Tolerance Test (50g 4-hours) — A 4-hour version of the oral glucose tolerance test where fasted patients (10hours overnight) consume a 50g of glucose solution & have glucose levels recorded up to every 5mins as well pancreatic and incretin responses at 10 fixed time points.
  Other Names: Modified OGTT; 50g OGTT
Drug: Matched isoglycemic clamp — A glucose drip will be infused at a variable rate that recreates the individual subjects blood glucose values obtained during their 4-hour modified oral glucose tolerance test. This test will therefore last 4-hours and again subjects will be fasted (10hours overnight) at the time of the test. The same blood tests will be performed at the same time points as the modified glucose tolerance test
  Other Names: isoglycemic clamp
Drug: Hyperglycemic clamp with concurrent GLP-1 infusion — An intravenous glucose infusion will be infused at a rate that maintains blood glucose at a level of 180-216mg/dL (10-12 mmol/l) (hyperglycemic clamp). After 60mins an infusion of GLP-1 will be commenced at a rate of 0.25pmol/kg/min for 60mins and then continued at a rate of 1.2pmol/kg/min for a further 60mins. Subjects will be blinded to what infusion they are receiving.
  Other Names: Glucagon-like peptide-1
Drug: Hyperglycemic Clamp with concurrent GIP infusion — An intravenous glucose infusion will be infused at a rate that maintains blood glucose at a level of 180-216mg/dL (10-12 mmol/l) (hyperglycemic clamp). After 60mins an infusion of GIP will be commenced at a rate of 1pmol/kg/min for 60mins and then continued at a rate of 4pmol/kg/min for a further 60mins. Subjects will be blinded to what infusion they are receiving.
  Other Names: gastric inhibitory polypeptide; glucose-dependent insulinotropic peptide
Drug: Hyperglycemic clamp with placebo infusion — An intravenous glucose infusion will be infused at a rate that maintains blood glucose at a level of 180-216mg/dL (10-12 mmol/l) (hyperglycemic clamp).
  After 60mins an infusion of normal saline will be commenced as a placebo infusion. It will be infused at a rate so that the total volume of fluid is similar to that infused during the other two hyperglycemic clamp interventions. Subjects will be blinded to what infusion they are receiving.
  Other Names: Hyperglycemic clamp with normal saline (0.9%) infusion
Other: Liquid Meal Test (Carbohydrate-rich) — A standardised liquid meal (carbohydrate-rich) containing approximately 500kcal would be administered to patients who had fasted overnight (10hrs). Over the next 4hours bloods would be sampled at 10 fixed time points to measure features of the incretin response to this type of meal.
Other: Liquid Meal Test (Fat-rich) — A standardised liquid meal (fat-rich) containing approximately 500kcal would be administered to patients who had fasted overnight (10hrs). Over the next 4hours bloods would be sampled at 10 fixed time points to measure features of the incretin response to this type of meal.
Other: Liquid Meal Test (Mixed) — A standardised liquid meal (mixed) containing approximately 500kcal would be administered to patients who had fasted overnight (10hrs). Over the next 4hours bloods would be sampled at 10 fixed time points to measure features of the incretin response to this type of meal.
Device: Continuous Glucose Monitoring — Continuous glucose monitoring entails wearing a small portable device, usually on the upper arm, for a period of three days. The device uses a small plastic tube to record the glucose level from interstitial fluid & every minute wirelessly transmits this information to a base unit to enable a very accurate estimate of average blood sugar control to be defined.
  Other Names: CGM; CGMS
  Groups: Cystic Fibrosis

SUMMARY:
Most Cystic fibrosis (CF) patients now commonly live well into adulthood, this means they are progressively accumulating damage to the insulin-secreting cells inside their pancreas. This explains why most adult patients have some degree of abnormal sugar regulation & rates of diabetes rise significantly with age. CF related diabetes is categorically different from other types of diabetes & its development is serious as it heralds a faster decline in lung function & a reduced life expectancy.

The hallmark of abnormal sugar handling in CF is high glucose levels after meals as the damaged pancreas responds abnormally slowly. Over 70% of the initial response of a healthy pancreas is induced, not by glucose alone, but by hormones released from the bowel known as incretins. We want to establish whether incretins are important in blood sugar handling in CF as specific drugs that enhance their effect are now available.

The study hypothesis is that the incretin system will function normally in patients with Cystic Fibrosis. To show this we will measure how much insulin secretion is dependant on incretin hormones in CF patients by comparing levels after a sugary drink test and then an intravenous glucose drip test (run at a rate that mimics the blood sugar levels obtained during the first test to make it a fair comparison ) - as incretins will only be produced in the first test when the sugar passes through the bowel any extra insulin produced will be due to these hormones. To detect resistance to the incretin hormones we will separately measure responses to direct infusions of the hormones themselves. We will explore which components of meals cause incretin hormone release from the bowel wall by measuring blood levels after different types of meals are consumed. Finally we will measure levels of the enzyme that breaks down the incretin hormones (DPP-4) to know if they are deactivated more quickly in people with CF. By describing the incretin system in CF we will considerably improve our understanding of this important condition as well as potentially highlighting new ways to treat it.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis as diagnosed by EITHER Cystic fibrosis transmembrane conductance regulator (CFTR) mutation on genotyping OR Positive sweat test (Chloride ≥60mmol/L after pilocarpine iontophoresis) AND Clinical features in keeping with a diagnosis of Cystic Fibrosis
* Clinically stable for at least 4 weeks without inpatient or outpatient treatment for an infective exacerbation - including antibiotics (other than long-term prophylactic therapy) or steroids

Exclusion Criteria:

* Active Pregnancy or <12 months Post-partum
* Clinically unstable patients
* Patients on long-term steroids
* Patients with known gastroparesis or previous surgery to the gastrointestinal tract (including vagotomy)
* History of organ transplant or planned organ transplant awaited
* Non-CF related diabetes (e.g. Type 1 or 2 Diabetes Mellitus)
* Active malignancy
* Clinically significant derangements in haematological or biochemical indices
* Clinical symptoms of malabsorption (frequent bowel motions/passing of undigested foodstuffs or steatorrhoea)
* Known difficult venous access
* Use of bile acid sequestrants in the previous 4 weeks

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The CF Cohort will be recruited from the population of Patients attending Adult CF Service at Liverpool Heart & Chest Hospital, Liverpool, United Kingdom
  The control group will be invited to participate from the general public. We will advertise our study through the Liverpool Heart & Chest Hospital and also via GP surgeries (Primary care clinics) in both electronic & paper forms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of Insulin & C-peptide secretion during a matched isoglycemic clamp | 4 hours
  Differences in Insulin & C-peptide secretion will be measured over a 4-hour period following an oral glucose tolerance test and then separately over the same period during a matched isoglycemic glucose infusion (which will recreate the glucose values obtained during the oral glucose tolerance test). The difference in these values can be wholly attributed to the effect of incretin hormones.
Volume of intravenous glucose required to maintain a hyperglycemic clamp at 180-216mg/dL | 3 hours
  A hyperglycemic clamp uses an intravenous glucose infusion to fix blood sugar at a certain level. We will use such a technique to fix blood sugar levels at 180-216mg/dL (10-12 mmol/l) for one hour then infuse either an incretin hormone (GLP-1/GIP) or placebo (sodium chloride) for a further two hours. The excess volume of intravenous glucose required during the last two hours of the test (compared to the first) will allow us to calculate what if any effect the incretin hormones have on the pancreas in patients with Cystic Fibrosis

SECONDARY OUTCOMES:
Serum DPP-4 levels | 0 mins
  We will measure serum DPP-4 levels on 2 separate occasions in both CF and control groups to establish if there are any differences in how rapidly the incretin hormones are deactivated between the groups
AUC incretin hormone levels (GLP-1/GIP) | 4 hours
  Incretin hormone levels (GLP-1/GIP) will be measured in response to an oral glucose tolerance test, an intravenous isoglycemic glucose infusion as well as in response to standardised meals of different composition (fat-rich, carbohydrate rich & mixed).

CONTACTS AND LOCATIONS:
Overall Officials: Gareth H Jones, MBChB, Principal Investigator — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom

REFERENCES:
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Mohan K, Miller H, Dyce P, Grainger R, Hughes R, Vora J, Ledson M, Walshaw M. Mechanisms of glucose intolerance in cystic fibrosis. Diabet Med. 2009 Jun;26(6):582-8. doi: 10.1111/j.1464-5491.2009.02738.x. PMID 19538232
- [Background] Milla CE, Warwick WJ, Moran A. Trends in pulmonary function in patients with cystic fibrosis correlate with the degree of glucose intolerance at baseline. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):891-5. doi: 10.1164/ajrccm.162.3.9904075. PMID 10988101
- [Background] Hameed S, Morton JR, Jaffe A, Field PI, Belessis Y, Yoong T, Katz T, Verge CF. Early glucose abnormalities in cystic fibrosis are preceded by poor weight gain. Diabetes Care. 2010 Feb;33(2):221-6. doi: 10.2337/dc09-1492. Epub 2009 Nov 12. PMID 19910502
- [Background] Dobson L, Sheldon CD, Hattersley AT. Validation of interstitial fluid continuous glucose monitoring in cystic fibrosis. Diabetes Care. 2003 Jun;26(6):1940-1. doi: 10.2337/diacare.26.6.1940-a. No abstract available. PMID 12766139
- [Background] Costa M, Potvin S, Hammana I, Malet A, Berthiaume Y, Jeanneret A, Lavoie A, Levesque R, Perrier J, Poisson D, Karelis AD, Chiasson JL, Rabasa-Lhoret R. Increased glucose excursion in cystic fibrosis and its association with a worse clinical status. J Cyst Fibros. 2007 Nov 30;6(6):376-83. doi: 10.1016/j.jcf.2007.02.005. Epub 2007 Apr 3. PMID 17409029
- [Background] Hillman M, Eriksson L, Mared L, Helgesson K, Landin-Olsson M. Reduced levels of active GLP-1 in patients with cystic fibrosis with and without diabetes mellitus. J Cyst Fibros. 2012 Mar;11(2):144-9. doi: 10.1016/j.jcf.2011.11.001. Epub 2011 Dec 3. PMID 22138561
- [Background] Anzeneder L, Kircher F, Feghelm N, Fischer R, Seissler J. Kinetics of insulin secretion and glucose intolerance in adult patients with cystic fibrosis. Horm Metab Res. 2011 May;43(5):355-60. doi: 10.1055/s-0031-1275270. Epub 2011 Mar 29. PMID 21448848
- [Background] Lanng S, Thorsteinsson B, Roder ME, Orskov C, Holst JJ, Nerup J, Koch C. Pancreas and gut hormone responses to oral glucose and intravenous glucagon in cystic fibrosis patients with normal, impaired, and diabetic glucose tolerance. Acta Endocrinol (Copenh). 1993 Mar;128(3):207-14. doi: 10.1530/acta.0.1280207. PMID 8480468